CLINICAL TRIAL: NCT01804530
Title: A Phase 1 Study to Assess Safety, Pharmacokinetics, and Pharmacodynamics of PLX7486 as a Single Agent in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Study of PLX7486 as Single Agent in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinued
Sponsor: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX119-01
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Solid Tumor; Tumors of Any Histology With Activating Trk (NTRK) Point or NTRK Fusion Mutations; Tenosynovial Giant Cell Tumor
Keywords: solid tumors; activating NTRK point or fusion mutations; Tenosynovial giant cell tumor; TGCT
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLX7486-TsOH, Dose escalation and RP2D (Experimental): Part 1: Open-label, sequential PLX7486-TsOH single-agent dose escalation in approximately 60 patients with solid tumors.
  Interventions: Drug: PLX7486 TsOH

INTERVENTIONS:
Drug: PLX7486 TsOH — PLX7486 TsOH capsules, 50mg

SUMMARY:
The objective of this study is to determine the safety, pharmacokinetics, maximum tolerated dose/recommended Phase 2 dose, and efficacy of PLX7486.

DETAILED DESCRIPTION:
Part 1. Open-label, sequential PLX7486 TsOH single-agent dose escalation in approximately 60 patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria

* Male or female ≥18 years old
* Patients with histologically confirmed solid tumors who:

  o Part 1: have tumor progression following standard therapy, have treatment-refractory disease, or for whom there is no effective standard of therapy
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiation of dosing and must agree to use an acceptable method of birth control. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year. Fertile men must also agree to use an acceptable method of birth control while on study drug and up to 3 months after the last dose of study drug.
* All associated toxicity from previous or concurrent cancer therapy must be resolved (to ≤Grade 1 or Baseline) prior to study treatment administration
* Patients with stable, treated brain metastases are eligible for this trial. However, patients must not have required steroid treatment for their brain metastases within 30 days of Screening.
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements
* Karnofsky performance status ≥70%
* Life expectancy ≥3 months
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria

* Other than the primary malignancy, active cancer (either concurrent or within the last 3 years) that requires non-surgical therapy (e.g., chemotherapy or radiation therapy), with the exception of surgically treated basal or squamous cell carcinoma of the skin, melanoma in situ, or carcinoma in-situ of the cervix
* Chemotherapy within 28 days prior to C1D1
* Biological therapy within 5 half-lives prior to C1D1
* Radiation therapy within 28 days or 5 half-lives prior to C1D1, whichever is longer
* Investigational drug use within 28 days or 5 half-lives, whichever is longer, prior to C1D1
* Part 1 only: (a) Patients with active or a history of glucose intolerance or diabetes mellitus and (b) Hemoglobin A1c ≥7%
* ≥Grade 2 sensory neuropathy at baseline
* Uncontrolled intercurrent illness (i.e., active infection) or concurrent condition that, in the opinion of the Investigator, would interfere with the study endpoints or the patient's ability to participate
* Refractory nausea and vomiting, malabsorption, small bowel resection that, in the opinion of the Investigator, would preclude adequate absorption
* Mean QTcF ≥450 msec (for males) or ≥470 msec (for females) at Screening
* The presence of a medical or psychiatric condition that, in the opinion of the Principal Investigator, makes the patient inappropriate for inclusion in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-08; Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Safety of PLX7486 as single agent as measured by adverse events and serious adverse events. | 1 year
Area under the plasma concentration-time curve [AUC0-t, AUC0-inf] | 1 year
  Area under the plasma concentration-time curve [AUC0-t, AUC0-inf] will be used to assess the pharmacokinetic profile of PLX7486.
Peak concentration (Cmax) | 1 year
  Peak concentration (Cmax) will be used to assess the pharmacokinetic profile of PLX7486.
Time to peak concentration (Tmax) | 1 year
  Time to peak concentration (Tmax) will be used to assess the pharmacokinetic profile of PLX7486.
Half life (t1/2) | 1 year
  Half life (t1/2) will be used to assess the pharmacokinetic profile of PLX7486.
Terminal elimination rate constant (Kel) | 1 year
  Terminal elimination rate constant (Kel) will be used to assess the pharmacokinetic profile of PLX7486.

SECONDARY OUTCOMES:
Duration of response (DOR) | 1 year
  Duration of response is defined as the number of days from the date of initial response (PR or better) to the date of first documented disease progression/relapse or death, whichever occurs first.
Progression-Free Survival (PFS) | 6 month
  Progression-free survival (PFS) is defined as the number of days from start of therapy to the date of documented disease progression/relapse, whichever occurs first.
Overall Response Rate (ORR) | 1year
Overall Survival (OS) | 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - John Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Medical University of South Carolina, Charleston, South Carolina